CLINICAL TRIAL: NCT04846907
Title: Mental Health and Emotional Aspects of Professionals Working in Pediatric Intensive Care Units During the COVID-19 Pandemic
Brief Title: Mental Health of Professionals Working in Pediatric Intensive Care Units During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Other Study IDs: COVID-EMOTION
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Covid19; Burnout, Professional; Stress Disorders, Post-Traumatic; Anxiety; Depression; Compassion Fatigue
Keywords: Covid19; Burnout; Post-Traumatic Stress Disorder; Anxiety; Depression; Compassion Fatigue
MeSH Terms: conditions — COVID-19; Burnout, Professional; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Compassion Fatigue; Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare personnel working in pediatric intensive care units during COVID-19 pandemic: Physicians, registered nurses, nurse technicians, physical therapists and other professionals; on duty, routine staff or fellow/residents working in participants PICU
  Interventions: Other: Web-based survey

INTERVENTIONS:
Other: Web-based survey — Eligible participants received emails or text messages with links to a REDCap-created and managed web-based questionnaire

SUMMARY:
Health professionals are extremely exposed to psychosocial risks, as they experience, in general, high levels of stress, anxiety, fatigue and suffering, due to the nature and location of their work. As a result, the health and well being of these professionals can be significantly compromised. In outbreaks of serious infectious diseases and pandemics, these risks become amplified and the health team is at greater risk of falling ill, presenting changes in mental health and psychological trauma, while caring for infected patients and becoming potential contaminants in their family and community.

The objective is to study the mental health of professionals who work in Pediatric Intensive Care Units (PICUs) in Brazil, during and after the COVID-19 pandemic. The primary outcome will be the prevalence of burnout in the team involved with the care of critically ill children. Secondary outcomes such as anxiety, depression, quality of professional life, compassionate fatigue and post-traumatic stress disorder will be measured. Possible associations between demographic, work and coping variables (social support and resilience) with mental and emotional health outcomes will be investigated, in an exploratory character.

It is a multicenter, observational, longitudinal study, with a descriptive and exploratory analytical component. Data collection will be carried out through an electronic survey during and after the COVID-19 pandemic.

DETAILED DESCRIPTION:
Health professionals are extremely exposed to psychosocial risks, as they experience, in general, high levels of stress, anxiety, fatigue and suffering, due to the nature and location of their work. As a result, the health and well being of these professionals can be significantly compromised. In outbreaks of serious infectious diseases and pandemics, these risks become amplified and the health team is at greater risk of falling ill, presenting changes in mental health and psychological trauma, while caring for infected patients and becoming potential contaminants in their family and community.

The objective is to study the mental health of professionals who work in Pediatric Intensive Care Units (PICUs) in Brazil, during and after the COVID-19 pandemic. The primary outcome will be the incidence of burnout in the team involved with the care of critically ill children. Secondary outcomes such as anxiety, depression, quality of professional life, compassionate fatigue and post-traumatic stress disorder will be measured. Possible associations between demographic, work and coping variables (social support and resilience) with mental and emotional health outcomes will be investigated, in an exploratory character.

It is a multicenter, observational, longitudinal study, with a descriptive and exploratory analytical component. Data collection will be carried out through an electronic survey during and after the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants that signed informed consent form

Exclusion Criteria:

* Refused to sign informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians, registered nurses, nurse technicians, physical therapists and other professionals; on duty, routine staff or fellow/residents working in participants PICU
Sampling Method: Non-Probability Sample
Enrollment: 1148 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of burnout as measured by Maslach Burnout Inventory (MBI) | Baseline
  Proportion of participants positive for Burnout as measured by MBI (Maslach et al), a self-report standardized 22-item questionnaire covering 3 domains: emotional exhaustion (EE), depersonalization (DP) and personal accomplishment (PA). Each subscale includes Likert-scaled questions ranging from 0 (never) to 6 (every day). Higher EE and DP scores and lower PA scores, more severe Burnout. Further analysis will be done to evaluate associations between Burnout presence and severity and demographic and laboral characteristics.

SECONDARY OUTCOMES:
Prevalence of anxiety as measured by Hospital Anxiety and Depression Scale (HADS) | Baseline
  Proportion of participants positive for anxiety as measured by HADS (Zigmond and Snaith), a self-report standardized 14-item questionnaire covering 1 anxiety 7-question subscale and 1 depression 7-question subscale. Each subscale includes Likert-scaled questions ranging from 0 to 3. Presence of anxiety symptoms when 9 or more points on anxiety subscale. Further analysis will be done to evaluate associations between anxiety presence and severity and demographic and laboral characteristics.
Prevalence of depression as measured by Hospital Anxiety and Depression Scale (HADS) | Baseline
  Proportion of participants positive for depression as measured by HADS (Zigmond and Snaith), a self-report standardized 14-item questionnaire covering 1 anxiety 7-question subscale and 1 depression 7-question subscale. Each subscale includes Likert-scaled questions ranging from 0 to 3. Presence of depression symptoms when 9 or more points on depression subscale. Further analysis will be done to evaluate associations between depression presence and severity and demographic and laboral characteristics.
Prevalence of Post-traumatic Stress Disorder (PTSD) as measured by PTSD Checklist DSM-5 (PCL-5) | Baseline
  Proportion of participants positive for PTSD as measured by PCL-5 (Weathers et al), a self-report standardized 20-item questionnaire covering 4 dimensions of symptoms: intrusions, avoidance, negative alterations in cognitions and mood and alterations in arousal and reactivity. Each subscale includes Likert-scaled questions ranging from 0 (not at all) to 4 (extremely). Presence of PTSD symptoms when 33 or more total points or positivity in each dimension. Further analysis will be done to evaluate associations between PTSD presence and severity and demographic and laboral characteristics.
Prevalence of Compassion Fatigue as measured by Professional Quality of Life 5 (ProQOL 5) scale | Baseline
  Proportion of participants positive for compassion fatigue and satisfaction as measured by ProQOL 5 scale (Stamm), a self-report standardized 30-item questionnaire covering 3 domains: compassion satisfaction (CS), Burnout (BO), secondary traumatic stress (ST). Each subscale includes Likert-scaled questions ranging from 1 (never) to 5 (very often). Scores are scaled between low (22 or less points), moderate (23 to 41) and high (42 or more) levels in each domain. Further analysis will be done to evaluate associations between CS, BO and ST presence and severity and demographic and laboral characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda L Setta, Principal Investigator — D'Or Institute for Research and Education
Locations (1):
- D'Or Institute for Research and Education, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oh N, Hong N, Ryu DH, Bae SG, Kam S, Kim KY. Exploring Nursing Intention, Stress, and Professionalism in Response to Infectious Disease Emergencies: The Experience of Local Public Hospital Nurses During the 2015 MERS Outbreak in South Korea. Asian Nurs Res (Korean Soc Nurs Sci). 2017 Sep;11(3):230-236. doi: 10.1016/j.anr.2017.08.005. Epub 2017 Aug 21. PMID 28991605
- [Background] Almutairi AF, Adlan AA, Balkhy HH, Abbas OA, Clark AM. "It feels like I'm the dirtiest person in the world.": Exploring the experiences of healthcare providers who survived MERS-CoV in Saudi Arabia. J Infect Public Health. 2018 Mar-Apr;11(2):187-191. doi: 10.1016/j.jiph.2017.06.011. Epub 2017 Jul 1. PMID 28676285
- [Background] Roy D, Tripathy S, Kar SK, Sharma N, Verma SK, Kaushal V. Study of knowledge, attitude, anxiety & perceived mental healthcare need in Indian population during COVID-19 pandemic. Asian J Psychiatr. 2020 Jun;51:102083. doi: 10.1016/j.ajp.2020.102083. Epub 2020 Apr 8. PMID 32283510
- [Background] Chan AO, Huak CY. Psychological impact of the 2003 severe acute respiratory syndrome outbreak on health care workers in a medium size regional general hospital in Singapore. Occup Med (Lond). 2004 May;54(3):190-6. doi: 10.1093/occmed/kqh027. PMID 15133143
- [Background] Greenberg N, Docherty M, Gnanapragasam S, Wessely S. Managing mental health challenges faced by healthcare workers during covid-19 pandemic. BMJ. 2020 Mar 26;368:m1211. doi: 10.1136/bmj.m1211. No abstract available. PMID 32217624
- [Background] Chen Q, Liang M, Li Y, Guo J, Fei D, Wang L, He L, Sheng C, Cai Y, Li X, Wang J, Zhang Z. Mental health care for medical staff in China during the COVID-19 outbreak. Lancet Psychiatry. 2020 Apr;7(4):e15-e16. doi: 10.1016/S2215-0366(20)30078-X. Epub 2020 Feb 19. No abstract available. PMID 32085839
- [Background] Buckley L, Berta W, Cleverley K, Medeiros C, Widger K. What is known about paediatric nurse burnout: a scoping review. Hum Resour Health. 2020 Feb 11;18(1):9. doi: 10.1186/s12960-020-0451-8. PMID 32046721
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Background] Wu PE, Styra R, Gold WL. Mitigating the psychological effects of COVID-19 on health care workers. CMAJ. 2020 Apr 27;192(17):E459-E460. doi: 10.1503/cmaj.200519. Epub 2020 Apr 15. No abstract available. PMID 32295761